CLINICAL TRIAL: NCT03753412
Title: Prospective Observational Study Regarding the Determinants of Functional Disability and Quality of Life in Patients Recovering From Severe Acute Cardiac or Respiratory Failure Considered for Mechanical Cardiorespiratory Support (CLEVERER)
Brief Title: Recovery From ICUAW Following Severe Respiratory and Cardiac Failure
Acronym: CLEVERER
Status: Recruiting | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 012370 CLEVERER
Record Dates: First submitted 2018-06-05; First posted 2018-11-27 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Intensive Care Unit Syndrome; Intensive Care Neuropathy; Intensive Care (ICU) Myopathy; Acute Respiratory Distress Syndrome; Cardiac Failure; Respiratory Failure; Critical Illness Myopathy
Keywords: Extra Corporeal Membrane Oxygenation (ECMO); Intensive Care Unit Acquired Weakness (ICUAW); Critical Illness Polyneuromyopathy (CIPM); Ultrasound (US); Health Related Quality of Life (HRQoL)
MeSH Terms: conditions — Muscular Diseases; Respiratory Distress Syndrome; Heart Failure; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Muscle Biopsies will be taken for histology examination at the time of surgery if the patients are centrally cannulated. Blood samples will be collected at specific time points to assess for mediators and markers of oxidative stress injury (e.g. 8-isoprostane), inflammation (e.g. interleukin-6 and soluble tumour necrosis factor receptor) and injury to multiple organs will be quantified. Urine will be collected to assess albumin-creatinine ration (ACR). Vascular endothelial cells will be analysed for cell culture and profile.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICUAW ECMO group: The physical and psychological effects of ICUAW on patients receiving extracorporeal membrane oxygenation for severe cardiorespiratory failure will be observed. Physical function and HRQoL will be analysed and correlated with RFcsa. Additionally, biological markers will be used to understand molecular and genomic profiles.

SUMMARY:
To observe and identify determinants of recovery from intensive care unit-acquired weakness (ICUAW) following a severe cardiorespiratory failure requiring extra-corporeal membrane oxygenation (ECMO). Additionally, to discover the effects of ICUAW on physical function and health-related quality of life (HRQoL) after critical illness. CLEVERER is a clinical observational pilot study.

DETAILED DESCRIPTION:
To identify determinants of recovery from ICUAW and to discover the effects of ICUAW on physical function and health-related quality of life (HRQoL) after critical illness. This phenomenon has become more evident over recent years and still requires extensive research.

ICUAW is an umbrella term for more specifically polyneuropathy and myopathy. Recent research has found that 50% of patients undergoing elective cardiac surgery lose significant muscle mass (9.6% in the wasters group) within the first seven days. These patients are receiving relatively uncomplicated surgery yet still suffering from muscle breakdown, which cannot be described by inactivity alone. The investigators wish to observe ICUAW in a real-life context, however, where cases are always severe. ICUAW can lead to a significant increase in mortality and morbidity. Risk factors for ICUAW include neuromuscular blocking agents, hyperglycaemia, inactivity and sepsis. The correlation between a patient group with severe cardiorespiratory failure and patient-centred outcomes during recovery such as functional ability and health-related quality of life (HRQoL) has been little studied.

Severe cardiac and respiratory failure can both be supported by a mechanical cardio-respiratory support (MCS) including extra-corporeal membrane oxygenation (ECMO); therefore referral for this intervention can be used as a marker of the severest form of cardiorespiratory failure. Both conditions are associated with a high incidence of collateral multi-organ dysfunction and mortality; as well as long-term morbidity, loss of independence and reduced quality of life. Patients with acute cardiac and respiratory failure referred to St Bartholomew's hospital for consideration of MCS will be recruited by advice/guidance from a personal and professional consultee.

Rectus femoris cross-sectional area (RFcsa) will be measured by ultrasound during the first week of admission and at pre-determined time points. The RFcsa will be correlated with indices of muscle strength, physical function and HRQoL. The investigators will also take blood and urine samples on arrival and at pre-defined intervals during the patients' admission for circulating and respiratory markers of sepsis, oxidative stress and organ injury. A muscle biopsy will be taken from the operation field if the patient is centrally cannulated when initiating ECMO.

The primary Objective is to identify determinants of recovery from ICUAW and to discover the effects of ICUAW on physical function and health-related quality of life (HRQoL) after severe cardiorespiratory failure. Specifically, to observe the cross-sectional area of the Rectus Femoris (RFcsa) and correlate this with muscle strength and HRQoL during recovery. RFcsa, hand-held dynamometry, knee straightening dynamometry, Free Fat Mass Index, standing and lying vital capacity, MRC-SS sum score and short physical performance battery (SPPB) will be observed. Also, HRQoL will be measured using the reintegration to normal living index (RNLI), hospital and anxiety depression score (HADS)and the EQ-5D-5L (EuroQol research foundation). Additionally, we have composed a 10 item questionnaire to assess pre-morbid functional status. The primary endpoint will be once all these data are gathered and analysed.

The secondary aim is to understand the molecular and genomic profile of blood samples and the histology of the muscle biopsies. The objective will be supported with additional data from urine analysis (albumin-creatinine ratio) and vascular endothelial cells. The secondary endpoint will be once these data are collected and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Above the age of 18
* Adults with severe cardio-respiratory failure requiring ECMO.
* Adults who have had personal and professional consultees agree to enrol them in the trial.

Exclusion criteria:

* Previous Stroke
* Neuromuscular disease
* Malignancy
* Underlying neuromuscular disease
* paediatrics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with severe cardiac or respiratory failure requiring extra-corporeal membrane oxygenation with no pre-existing muscle weakness or wasting.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-04-09 (Actual); Primary Completion 2026-09-26 (Estimated); Study Completion 2026-09-26 (Estimated)

PRIMARY OUTCOMES:
To observe the change in cross sectional area of the Rectus Femoris (RFcsa, measured in cm2) during critical illness and recovery. | Up to approximately 1 year.
  RFcsa will be calculated using B-mode ultrasound (US) at pre-determined time points. Additionally, the images acquired will have histogram analysis in adobe photoshop software. The RFcsa will be correlated with indices of muscle strength and HRQoL. A larger RFcsa with reduced pixel density suggests greater muscle quality and function.
To Observe a change in Hand Held Dynamometry strength and correlate this with RFcsa, function and HRQoL during critical illness and recovery. | Up to approximately 1 year.
  Hand-held dynamometry will be calculated using the JAMAR hand-held hydraulic dynamometer. We will assess both hands and take the mean of 3 trials, producing a maximal grip result. A higher score indicates better global strength and function.
To observe a change in Knee straightening dynamometry, strength and joint moment (torque) and correlate this with RFcsa, function and HRQoL during critical illness and recovery. | Up to approximately 1 year
  The test will be conducted using a Lafayette Manual Muscle Tester. Joint knee moment (torque) and strength will be measured. A higher result from joint knee moment and strength indicates a greater global strength and function.
To test the Medical Research Council Sum Score (MRC-SS). MRC-SS measures global strength and ambulation | Up to approximately 1 year.
  This test will be conducted once to reaffirm whether patients' have ICUAW. A score can range from 0 (paralysis) to 60 (normal strength). A score of less than 48 indicates the patient has ICUAW. Therefore, a lower score is associated with worse outcomes.
To observe a change in Short Physical Performance Battery (SPPB) and correlate this with RFcsa, function and HRQoL during critical illness and recovery | Up to approximately 1 year.
  SPPB will be used as a further marker of functional status. The patient can score between 0 (poor functional status) and 12 (good functional status).
Lying and Standing Vital Capacity (FVC - forced vital capacity) and correlate this with RFcsa, function and HRQoL during critical illness and recovery. | Up to approximately 1 year
  Lying and standing vital capacity will be measured using a hand held spirometer. The test score will be compared to the predicted normal value based on age, height, race and gender. A result is considered normal if it is 80 percent or more of the predicted value.
To measure a change in Free Fat Mass Index (FFMI) and correlate this with RFcsa, function and HRQoL during critical illness and recovery. | Up to approximately 1 year
  Free fat mass index (FFMI) and free fat mass (FFM) will be measured using the bodystat 1500 device. Other values will also be recorded from the test including body fat percentage and lean mass percentage. The body stat 1500 is an electrical device that uses electrical impedance to obtain results (objective data). Results will be compared to predicted values based on age, sex, height and weight.
To measure the EQ-5D-5L (Euroscore) to assess general health and correlate this with the primary objective (RFcsa). | Up to approximately 1 year
  EQ5D-5L is a standardised tool that provides a simple generic measure of health. A summation of all the levels will be converted to a single index value using the EQ5D-5L crosswalk index value calculator. The general health score can range from 0 (worst health imaginable) to 100 (best health imaginable). Additionally, a health state ranging from level 1 (indicating no problem) to level 5 (indicating extreme problems) can be calculated using the descriptive system and its five dimensions.
Hospital anxiety and depression score (HADS) to assess HRQoL and correlate this with the overall primary objective (RFcsa). | Up to approximately 1 year
  The HADS is an assessment that measures whether a patient is suffering from anxiety or depression. HADS is a self assessment consisting of 16 items. A result between 0 and 7 indicates a normal case, between 8 and 10 indicates borderline abnormal and between 11 and 21 indicates abnormal levels of anxiety and depression.
Reintegration to normal living index (RNLI) to assess HRQoL and correlate this with the overall primary objective (RFcsa). | Up to approximately 1 year
  The RNLI is a 5 domain 11-tool item aimed at assessing the degree to which patients' who have experienced traumatic and incapacitating illness achieve reintegration into society. The RNLI score is based out of 110, which will be proportionally converted to create a score of 100. Zero indicates no integration whereas 100 implies full integration.
10-item questionnaire to assess HRQoL (pre-morbid functional status) and correlate this with the overall primary objective. | Day 0 (on admission)
  This is a locally devised questionnaire that is answered by the patients' next of kin due to them being incapacitated. We will correlate these results with the other HRQoL questionnaires.

SECONDARY OUTCOMES:
The secondary aim is to understand the molecular profile (bloods). | Up to approximately 1 year
  Blood analysis will contain and analyse but not limited to markers of oxidative stress injury, inflammation, MiRNA and injury to multiple organs will be quantified. We will collect, store and analyse buffy coat and plasma to understand these profiles.
Urine Analysis | Up to approximately 1 year
  Urine analysis measures albumin-creatinine ratio (ACR).
Muscle Biopsy | Intra operatively
  A muscle biopsy will be taken from patients whilst under anaesthesia. The biopsy observes pathways relevant to muscle homeostasis using biochemical and molecular techniques.
Vascular endothelial cell sampling | Day 0.
  Cell samples will be acquired from insertion of the central line.
Cardiac post operative morbidity score (C-POMS) will be used to calculate total morbidity risk. | Time Frame: Day 3, day 5, day 8 and day 15 post ECMO initiation.
  C-POMS is additional data that will be collected and analysed. C-POMS is a validated tool assessing in-hospital morbidity burden (score 0-13) derived by noting the presence of 13 morbidity domains (pulmonary, infectious, renal, gastrointestinal, cardiovascular, neurological, haematological, wounds, pain, endocrine, electrolytes, review and assisted ambulation) on days 3, 5, 8 and 15 after cardiac surgery. A higher score indicates a greater morbidity burden. Although ECMO is not considered cardiac surgery we can still utilise C-POMS as a descriptive measure.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Griffiths, PhD FRCP, Principal Investigator — Substantive Employee and primary supervisor to PhD student; Julie Sanders, MSc, PhD, Principal Investigator — Director of research and supervisor to PhD student; Ashley Thomas, MSc, Principal Investigator — Substantive employee and PhD student
Locations (1):
- St Bartholomew's hospital (Barts NHS trust), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bloch SA, Donaldson AV, Lewis A, Banya WA, Polkey MI, Griffiths MJ, Kemp PR. MiR-181a: a potential biomarker of acute muscle wasting following elective high-risk cardiothoracic surgery. Crit Care. 2015 Apr 7;19(1):147. doi: 10.1186/s13054-015-0853-5. PMID 25888214